CLINICAL TRIAL: NCT03302169
Title: Prospective Randomized Controlled Trial to Compare Early Urinary Continence Recovery After Robotic Assisted Radical Prostatectomy With or Without Posterior Rhabdosphincter Reconstruction.
Brief Title: Trial to Compare Urinary Continence Recovery After Robotic Radical Prostatectomy With or Without Rhabdosphincter Reconstruction.
Acronym: RHABDO-PROST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: PR(AG)330/2016
Record Dates: First submitted 2017-08-15; First posted 2017-10-05 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Urinary Incontinence
Keywords: Prostate Cancer; Urinary incontinence; Radical prostatectomy; Rhabdosphincter; Robotic Surgery
MeSH Terms: conditions — Urinary Incontinence; Prostatic Neoplasms | interventions — Posterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized controlled trial to assess early urinary continence recovery rates after robotic assisted radical prostatectomy when a posterior rhabdosphincter reconstruction is performed or not.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior Rhabdosphincter Reconstruction (Experimental): Patients in who posterior rhabdosphincter reconstruction is performed
  Interventions: Procedure: Radical prostatectomy with posterior rhabdosphincter reconstruction
- Standard Technique (Active Comparator): Patients in who posterior rhabdosphincter reconstruction is NOT performed, Standard technique.
  Interventions: Procedure: Radical prostatectomy without posterior rhabdosphincter reconstruction

INTERVENTIONS:
Procedure: Radical prostatectomy with posterior rhabdosphincter reconstruction — To suture the Denonvilliers fascia and bladder to the median dorsal raphe according to Rocco technique.
  Other Names: Rocco reconstruction technique; Posterior reconstruction; Rocco Stitch
  Arms: Posterior Rhabdosphincter Reconstruction
Procedure: Radical prostatectomy without posterior rhabdosphincter reconstruction — Standard technique with a running suture to perform the urethrovesical anastomosis
  Arms: Standard Technique

SUMMARY:
This is a prospective randomized controlled trail to assess early urinary continence recovery rates after robotic assisted radical prostatectomy when a posterior rhabdosphincter reconstruction is performed or not. A hundred forty-six patients with clinically localized and histological confirmed prostate cancer will be enrolled. Continence recovery is defined in the present study as declared urinary continence (absence of incontinence episodes) in the physician interview as no pad use. Continence rates will be explored also by EPIC, ICIQ-SF, IPSS questionnaires 1, 6 and 12 months after the procedure. The sexual function as the secondary objective will be assessed by SHIM questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of prostate cancer
* Localized or locally advanced prostate cancer
* Informed consent signed

Exclusion Criteria:

* Presence of urinary incontinence prior to the procedure
* Previous radiation therapy of the prostate or pelvis
* Presence of any prostatic surgery prior to the procedure
* Prior medical history of psychiatric diseases or drug addiction
* Any condition that contraindicates a radical prostatectomy

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Number of patients using 0-1 PAD/d (EPIC-26 question_5) at 1st monthNumber of patients using 0-1 PAD/d (EPIC-26 question_5) at 1st month | 1 month after surgery
  Absence of urinary incontinence (number of PADs/d)
Number of patients using 0-1 PAD/d (EPIC-26 question_5) at 6th month | 6 months after surgery
  Absence of urinary incontinence (number of PADs/d)

SECONDARY OUTCOMES:
early urinary recovery quantification in Grams (PAD-test 24h) | one day before catheter removal, 2 weeks before and 1 month before
  PAD-test during the first month after surgery
Number of patients using 0-1 PAD/d (EPIC-26 question_5) at 12th month | 12 months after surgery
  Absence of urinary incontinence (number of PADs/d)
Erectile function | 1, 6 and 12 months
  SHIM assessment
Quality of life I: urinary and bowel function | 1, 6 and 12 months
  EPIC-26 urinary and digestive function
Quality of life II: urinary function | 1, 6 and 12 months
  ICIQ-SF assessment of urinary function
Quality of life III: urinary function | 1, 6 and 12 months
  IPSS assessment of urinary function
Oncological outcome: Biochemical free-recurrence status | 1, 6 and 12 months
  serum PSA assessment. Biochemical free-recurrence status = PSA <0.2
Anatomopathological parameters: Surgical margins | 1 month
  Surgery margins in prostatectomy specimens
Anatomopathological parameters: pTNM classification | 1 month
  Pathological pTNM in prostatectomy specimens

CONTACTS AND LOCATIONS:
Overall Officials: Juan Morote, PhD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salazar A, Regis L, Planas J, Celma A, Trilla E, Morote J. Continence definition and prognostic factors for early urinary continence recovery in posterior rhabdosphincter reconstruction after robot-assisted radical prostatectomy. Post-hoc analysis of a randomised controlled trial. Actas Urol Esp (Engl Ed). 2022 Apr;46(3):159-166. doi: 10.1016/j.acuroe.2021.06.012. Epub 2022 Mar 7. English, Spanish. PMID 35272967
- [Derived] Salazar A, Regis L, Planas J, Celma A, Santamaria A, Trilla E, Morote J. A Randomised Controlled Trial to Assess the Benefit of Posterior Rhabdosphincter Reconstruction in Early Urinary Continence Recovery after Robot-assisted Radical Prostatectomy. Eur Urol Oncol. 2022 Aug;5(4):460-463. doi: 10.1016/j.euo.2021.02.005. Epub 2021 Feb 27. PMID 33653674